CLINICAL TRIAL: NCT05398016
Title: Testing a Task Sharing Model to Expand Access to Mental Health Services for Anxiety
Brief Title: Strategies for Treating Anxiety Research Study
Acronym: STARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNLV-2022-263
Record Dates: First submitted 2022-05-19; First posted 2022-05-31 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-03

CONDITIONS: Anxiety Disorders; Anxiety
Keywords: task sharing; task shifting; lay counselor; psychological treatment
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single arm pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-intensity behavioral intervention (Experimental): Brief behavioral intervention for mild-to-moderate symptoms of anxiety. Delivered via weekly sessions by a trained lay counselor ("coach").
  Interventions: Behavioral: low-intensity intervention for anxiety

INTERVENTIONS:
Behavioral: low-intensity intervention for anxiety — Brief (6-8 weekly 30-min sessions) delivery of a structured behavioral treatment for mild-to-moderate anxiety. Treatment will be based on principles of cognitive behavioral therapy (CBT).

SUMMARY:
This single-arm pilot clinical trial will evaluate the feasibility, acceptability, and engagement of target mechanism, and preliminary impact of a low-intensity behavioral intervention for mild-to-moderate anxiety disorders. Treatment will delivered by trained lay counselors ("coaches;" n = 5-6) to 2-5 patient participants each depending on enrollment and scheduling (n = up to 25).

DETAILED DESCRIPTION:
Anxiety is the most common adult mental health condition. Left untreated, it is costly and imparts significant personal and public health burden. Evidence-based psychotherapy (EBP) is an acceptable and effective first-line treatment; however, rural, low-income, and other underserved areas suffer from provider shortages, rendering such treatment largely unavailable. International contexts are beginning to address this problem using provider task sharing, in which low-intensity behavioral health services are delivered by non-specialist health workers (i.e., those with no prior training as a mental health professional). This approach is designed to improve access to care, particularly for those with mild-to-moderate symptoms, and free up limited expert resources. What is lacking is a brief, evidence-based, low-intensity behavioral intervention for mild-to-moderate anxiety disorders as well as an implementation blueprint (e.g., identifying appropriate clinical setting, stakeholder needs, supervision requirements, other counselor and clinic supports) needed to successfully implement and sustain such a novel service model in U.S. contexts. This study will begin to address the above problem in two phases, while creating the foundation for a longterm research program and external funding applications. The primary objective of this work is to develop and preliminarily test a brief intervention for anxiety appropriate for primary care and other non-specialty contexts. Investigators will test the intervention and delivery method via a small, single-arm pilot clinical trial. Non-specialists "coaches" will be trained undergraduate or post-baccalaureate student "coaches" (approx. 5-6 to accommodate patient participant scheduling), each working with three patient participants with anxiety (N = up to 25) to provide preliminary data on fidelity, feasibility, acceptability, preliminary clinical outcomes, and engagement of the target clinical mechanism of avoidance. The activities of these aims will develop community and clinical partnerships for testing and future implementation of low-intensity treatment paradigms.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years,
* score on Beck Anxiety Inventory (BAI) ≥ 16,
* ability to speak English
* willing and able to attend in-person study visits at UNLV
* community dwelling

Exclusion Criteria:

* other psychological conditions rendering the person unlikely to benefit from a brief treatment, including psychosis, bipolar disorder, cognitive impairment, and substance abuse or dependence (comorbid depression permitted);
* active suicidal ideation or intent;
* concurrent receipt of regular individual psychotherapy;
* use of anxiolytic medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenna Renn, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be shared with investigators whose proposed data use has been approved through requests to the Principal Investigator. These requests will be considered after publication of the main outcome paper from the project.
Supporting Information: Study Protocol, ICF
Time Frame: Upon publication of main outcomes paper; estimated Jan 2026; will remain available indefinitely
Access Criteria: Requirements:
  Scientific rationale: A strong justification for why the data is needed and how it will contribute to scientific advancement.
  Ethical considerations: A demonstration that the research plan is ethically sound and that potential risks to participants are minimized.
  Data security and privacy: Measures to ensure the confidentiality and security of the data.
  Commitment to responsible use: A pledge to use the data ethically and responsibly, in accordance with the study's protocol and relevant regulations.

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Participants: Low-intensity behavioral intervention: Brief behavioral intervention for mild-to-moderate symptoms of anxiety. Delivered via weekly sessions by a trained lay counselor ("coach").
- Coach Participants: Adults with advanced undergraduate standing or baccalaureate who complete required training and consent to serve as supervised coaches (nonspecialist providers), delivering the brief intervention to patient participants.
Period: Overall Study
Arm/Group | Patient Participants | Coach Participants
Started | 21 | 6
Completed | 17 | 6
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patient Participants: Adults (18+) with clinically elevated symptoms of anxiety who received brief behavioral intervention for mild-to-moderate symptoms of anxiety. Delivered via weekly sessions by a trained lay counselor ("coach").
- Coach Participants: Nonspecialists who were trained and supervised to deliver the experimental intervention with the patient participants. Referred to as "coaches."
- Total: Total of all reporting groups
Arm/Group | Patient Participants | Coach Participants | Total
Number analyzed (Participants) | 21 | 6 | 27
Age, Continuous [Mean (Full Range); unit: years] — Population: Age was collected and analyzed for patient participants only to characterize the sample. Age was not collected as a continuous variable for coach participants.
  years
    number analyzed (Participants) | 21 | 0 | 21
    (all) | 28.9 [19 to 42] |  | 28.9 [19 to 42]
Age, Customized [Count of Participants; unit: Participants] — Proportion of participants aged 18 and older
  Participants
    18 years of age or older | 21 | 6 | 27
Sex: Female, Male [Count of Participants; unit: Participants] — Data were collected as gender with multiple options. Population: Data were collected as gender with multiple options.
  Participants
    Female | 18 | 5 | 23
    Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 19 | 5 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 3 | 12
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: Participants]
  United States | 21 | 6 | 27
Generalized Anxiety Disorder (GAD-7) scale [Mean (Standard Deviation); unit: units on a scale] — The 7-item Generalized Anxiety Disorder scale (GAD-7) collects participant-reported anxiety symptom severity and frequency across seven symptoms (e.g., worry, psychosomatic symptoms). Items are score on a 4-point scale, 0=not at all to 3=nearly every day. Total summary scores range from 0-21, with higher scores indicating greater severity (worse) anxiety. This was only collected on patient participants. The GAD-7 was not collected from coach (interventionist) participants. Population: participant-reported anxiety symptom severity; only collected on patient participants
  units on a scale
    number analyzed (Participants) | 21 | 0 | 21
    (all) | 11.9 (2.8) |  | 11.9 (2.8)

OUTCOME MEASURES:

1. Secondary Outcome: Acceptability of Intervention Measure (AIM)
Description: Self-report measure assessing perceived acceptability of the intervention (an implementation outcome). Scores range from 4-20; higher scores indicate a higher degree of perceived acceptability. Completed by the trained lay counselors.
Time Frame: Post-implementation (up to 1 year)
Measure: Mean (Full Range); unit: scores on scale
Groups:
- Coach Participants: Nonspecialists who were trained and supervised to deliver the experimental behavioral intervention to patient participants.
Arm/Group | Coach Participants
Number analyzed (Participants) | 6
scores on scale | 4.88 [4 to 5]

2. Secondary Outcome: Feasibility of Intervention Measure (FIM)
Description: Self-report measure assessing perceived feasibility of the intervention (an implementation outcome). Scores range from 4-20; higher scores indicate a higher degree of perceived feasibility. Completed by the trained lay counselors.
Time Frame: Post-implementation (up to 1 year)
Measure: Mean (Full Range); unit: scores on scale
Arm/Group | Coach Participants
Number analyzed (Participants) | 6
scores on scale | 5 [5 to 5]

3. Secondary Outcome: Implementation Appropriateness Measure (IAM)
Description: Self-report measure assessing perceived appropriateness of the intervention (an implementation outcome). Scores range from 4-20; higher scores indicate a higher degree of perceived appropriateness. Completed by the trained lay counselors.
Time Frame: Post-implementation (up to 1 year)
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Coach Participants
Number analyzed (Participants) | 6
scores on a scale | 4.88 [4 to 5]

4. Primary Outcome: Number of Patient Participants Retained in the Intervention (Out of All of Those Enrolled), as Measured by Completion to All Study Treatment Visits.
Description: Retention of patient participants will be measured as an implementation outcome. This will entail quantifying the number of patients who complete the entire course of treatment out of all of those enrolled.
Time Frame: through treatment completion, up to 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Patient Participants: Adults (18 years and older) with elevated anxiety symptoms who received experimental intervention delivered by coach participants.
Arm/Group | Patient Participants
Number analyzed (Participants) | 21
Participants | 17

5. Primary Outcome: Change in Anxiety Symptoms
Description: (Patient outcome) Change between pre- and post-treatment will be assessed using the Structured Interview Guide for the Hamilton Anxiety Scale. This is a clinician-rated measure consisting of 14 items, each defined by a series of symptoms, to measure both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Total summary score ranges from 0 to 56, with higher scores indicating more severe and frequent symptoms of anxiety. A corresponding interview guide will be used to increase the reliability of the Hamilton Anxiety Scale. This measure has demonstrated sensitivity to change in clinical trials.
Time Frame: change in anxiety between pre- and post-treatment (6-8 weeks)
Population: per protocol analysis of completers (n = 17)
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Patient Participants
Number analyzed (Participants) | 17
scores on scale | 4.69 (4.44)

6. Primary Outcome: Change in Avoidance
Description: (Patient outcome) Change in avoidance will be measured using the Multidimensional Experiential Avoidance Questionnaire (MEAQ). This is a 62-item self report assessment of avoidance. Total scores range from 62 to 372; higher scores reflect higher levels of avoidance. This will be used to measure activation of target mechanism of avoidance.
Time Frame: change in avoidance between pre- and post-treatment (6-8 weeks)
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Patient Participants
Number analyzed (Participants) | 17
scores on scale | 6.68 (23.64)

7. Secondary Outcome: World Health Organization's Disability Assessment Schedule 2.0 (WHODAS 2.0)
Description: This 12-item generic health-status measure assesses functioning across six domains: communication, mobility, self-care, interpersonal, life activities, and participation. Each item is scored on a 5-point scale (0 = no difficulty to 4 = extreme difficulty or cannot do). The scores for each item are summed to create a total score. A total score is possible from 0-48, with 48 representing the highest level of disability.
Time Frame: change in functioning between pre- and post-treatment (6-8 weeks)
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Patient Participants: Patient participants received the experimental intervention
Arm/Group | Patient Participants
Number analyzed (Participants) | 17
score on a scale | 4.600 (10.99)

8. Primary Outcome: Sustained Change in Anxiety Symptoms
Description: (Patient outcome) Change in anxiety between baseline (pre-treatment) and follow-up (12 weeks; 6 week after intervention end) will be assessed using the Structured Interview Guide for the Hamilton Anxiety Scale. This is a clinician-rated measure consisting of 14 items, each defined by a series of symptoms, to measure both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Total summary score ranges from 0 to 56, with higher scores indicating more severe and frequent symptoms of anxiety. A corresponding interview guide will be used to increase the reliability of the Hamilton Anxiety Scale. This measure has demonstrated sensitivity to change in clinical trials.
Time Frame: change in anxiety between pre-treatment and follow-up (12 weeks)
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Patient Participants
Number analyzed (Participants) | 17
scores on scale | 4.75 (4.40)

9. Other Pre Specified Outcome: Sustained Change in Avoidance
Description: (Patient outcome) Sustained change in avoidance after treatment (12 weeks follow-up; this is 6 weeks after treatment end) will be measured using the Multidimensional Experiential Avoidance Questionnaire (MEAQ). This is a 62-item self report assessment of avoidance. Total scores range from 62 to 372; higher scores reflect higher levels of avoidance. This will be used to measure activation of target mechanism of avoidance.
Time Frame: change in avoidance between pre-treatment and follow-up (12 weeks)
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: scores on scale
Groups:
- Patient Participants: patient participants who received experimental treatment
Arm/Group | Patient Participants
Number analyzed (Participants) | 17
scores on scale | 11.71 (10.93)

ADVERSE EVENTS:
Time Frame: Active treatment (6-8 weeks)
Description: Patient participants were non-systematically assessed for adverse events, such as self-reporting in treatment sessions or as follow-up questions if they self-reported such information in routine assessments. Coach participants were non-systematically assessed for serious adverse events in weekly coach supervision meetings, such as self-reporting.
Arm/Group | Patient Participants | Coach Participants
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/6
Other Adverse Events (participants affected / at risk) | 0/21 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT05398016/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT05398016/SAP_001.pdf